CLINICAL TRIAL: NCT05937503
Title: Efficiency of Manual Therapy on Central Sensitization in Patients With Nonspecific Chronic Back Pain.A Randomized Controlled Study.
Brief Title: Efficiency of Manual Therapy on Central Sensitization in Patients With Nonspecific Chronic Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, NAİME ULUG, PhD., Atılım University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-59394181-604.01.02-33380
Record Dates: First submitted 2023-06-27; First posted 2023-07-10 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Central Sensitization; Manual Therapy
Keywords: central sensitization; manual therapy; non-specific low back pain
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled study
Who Masked: Participant
Masking Description: Participant will not informed about the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy (Experimental): Manual therapy group
  Interventions: Other: manual therapy; Other: conventional physiotherapy
- Conventional physiotherapy (Other): Conventional physiotherapy group
  Interventions: Other: manual therapy; Other: conventional physiotherapy

INTERVENTIONS:
Other: manual therapy — The manual therapy group will receive a 4-week manual therapy plus conventionel physiotherapy.
  Other Names: conventional physiotherapy
Other: conventional physiotherapy — Control group will only receive conventionel physiotherapy intervention.

SUMMARY:
Central sensitization (CS) is defined as the increased responsiveness of nociceptive neurons in the central nervous system to normal or subthreshold afferent input. CS has been proposed as an underlying mechanism of chronic pain in musculoskeletal disorders including low back pain (LBP).

The aim of this study is to investigate the effect of manual therapy on central sensitization in patients with nonspecific chronic LBP.

DETAILED DESCRIPTION:
A total of 40 LBP patients aged between 24-64 with CSS will be randomized into two groups. The manual therapy group will receive a 4-week manual therapy (two sessions/week) plus the conventional physiotherapy program, while the control group will only receive conventional physiotherapy. Before and after the interventions pain intensity (VAS), and scores of three questionnaires: Oswestry Disability Index (ODI), Central Sensitization Inventory (CSI), and the 36-item Short Form Health Survey Questionnaire (SF-36) will be recorded.The outcomes of the study will be analyzed by appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* non-spesific low back pain patients with pain longer than 12 weeks
* aged between 20-64 years male and female participants

Exclusion Criteria:

* concomitant disease that would interfere with treatment
* pregnancy
* have had any spinal surgery or fracture

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-17 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Up to one month
  A 10 cm Visual Analog Scale will be used to determine the severity of pain, with numbers ranging from "0" (no pain) to "10" (unbearable pain)
Central Sensitization | Up to one month
  Central Sensitization Inventory (CSI) scale will be used severity of central sensitization.The total score range of the scale, which consists of a total of 25 questions, is between 0-100 points. Central sensitization with a score of 40 and above is considered positive. An increase in the total score indicates an increase in the level of central sensitization.

SECONDARY OUTCOMES:
Oswestry Disability Index | Up to one month
  Oswestry Disability Index (ODI) will be used to measure disability level
Health Survey | Up to one month
  36-item Short Form Health Survey Questionnaire (SF-36) will be used
Hospital Anxeity and depresssion | Up to one month
  Hospital Anxeity and Depression Scale will be used. The cut-off points for caseness of anxiety or depression is 8/21 for anxiety or depression. For anxiety (HADS-A) this gave a specificity of 0.78 and a sensitivity of 0.9. For depression (HADS-D) this gave a specificity of 0.79 and a sensitivity of 0.83.
  The scores of the scale are as follows: 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Naime Ulug, Ankara, Select State
  - Atılım University, Ankara

IPD SHARING:
Plan to Share IPD: No